CLINICAL TRIAL: NCT06267287
Title: Microbiological Structure of Pathogens of Periprosthetic Infection of Large Joints in the Post-Covid Period
Status: Completed | Type: Observational
Sponsor: Federal State Budgetary Organization, Federal Center for Traumatology, Orthopedics and Arthroplasty (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-4
Record Dates: First submitted 2024-01-24; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-01

CONDITIONS: Joint Infection; Periprosthetic Left Knee Joint Infection
Keywords: periprosthetic infection; antibiotic resistance; Staphylococcus epidermidis; pathogens of periprosthetic infection; COVID-19; empirical antibiotic therapy
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cases of PJI 2018-2019: All cases of monomicrobial and polymicrobial periprocthetic infection for 2018-2019. Microbiological identification of pathogens of periprosthetic infections and determination of their sensitivity to antibiotics.
  Interventions: Diagnostic Test: Microbiological examination of the patient's biological material and determination of antibiotic resistance
- cases of PJI 2021-2022: All cases of monomicrobial and polymicrobial periprocthetic infection for 2021-2022. Microbiological identification of pathogens of periprosthetic infections and determination of their sensitivity to antibiotics.
  Interventions: Diagnostic Test: Microbiological examination of the patient's biological material and determination of antibiotic resistance

INTERVENTIONS:
Diagnostic Test: Microbiological examination of the patient's biological material and determination of antibiotic resistance — Isolated microorganisms were identified based on growth in one or more cultures obtained from punctate synovial fluid, intraoperative tissues, and from removed implants (after their ultrasonic treatment). At least 4 samples of intraoperative material (tissue biopsies, joint aspirate, removed endoprosthesis components) were taken from patients for examination. The endoprosthesis components removed during surgery were placed in a sterile plastic container and delivered to the laboratory. In the laboratory, saline solution was added to the container and processed in an ultrasonic machine according to the author's method. Identification of isolated microorganisms and sensitivity to antibiotics was carried out using an automatic analyzer and a semi-automatic analyzer using kits, test systems. Sensitivity to antibacterial drugs was tested using the disk diffusion method and analyzer kits. Antibiotic sensitivity assessment was carried out in accordance with the criteria of EUCAST.
  Other Names: Identification of the infectious agent and determination of antibiotic resistance

SUMMARY:
Background. Infection is the most common complication of complications after joint arthroplasty. During the COVID-19 pandemic increased used antibacterial drugs by adults, this could change the spectrum of infectious agents and their antimicrobial resistance. The purpose of the study is to evaluate the microbial diversity of pathogens of periprosthetic infection in the pre- and post-Covid period, determining the sensitivity of the leading pathogens to antibiotics. Materials and methods. A comprehensive comparative retrospective study was carried out on 342 cases of monomicrobial and polymicrobial periprosthetic infection (PPI) of limb joints with microbiological growth of microorganisms in the pre-Covid (2018-2019) and post-Covid (2021-2022) periods.

DETAILED DESCRIPTION:
A continuous comparative retrospective study of cases of PJI of the joints of the extremities with positive microbiological growth of microorganisms in the pre-Covid (2018-2019) and post-Covid (2021-2022) periods was carried out on the data basis from the medical information system (MIS) of the Federal Center for Traumatology, Orthopedics and Arthroplasty of Ministry of Health of Russia (Cheboksary, Russia), hereinafter referred to as the Center.

Verification of the diagnosis of deep PJI was carried out according to the diagnostic criteria of the Society for Musculoskeletal Infections.

The sample included cases of deep and superficial infection after arthroplasty of the knee, hip, shoulder and wrist joints, regardless of the location of the primary operation. Isolated microorganisms were identified based on growth in one or more cultures obtained from punctate synovial fluid, intraoperative tissues, and from removed implants (after their ultrasonic treatment).

The infection was classified as polymicrobial or monomicrobial. The role of the leading pathogen was determined in the structure of monomicrobial infection. Polymicrobial infection is represented by cases of simultaneous isolation of two or more pathogens in one patient. The antibiotic resistance profile included all isolated pathogens of mono- and polymicrobial PJI.

At least 4 samples of intraoperative material (tissue biopsies, joint aspirate, removed endoprosthesis components) were taken from patients for examination.

The aspirate from the joint was placed into FA plus, FN plus bottles of the Bact/Alert 3D analyzer (Bio Merieux, France). If the sample volume was insufficient (less than 1 ml), it was inoculated into a vial with Schedler's broth and, when turbid, subcultured onto solid media.

The endoprosthesis components removed during surgery were placed in a sterile plastic container and delivered to the laboratory. In the laboratory, saline solution was added to the container and processed in an ultrasonic machine according to the author's method. After ultrasonication, 0.5 ml of the resulting liquid was applied to solid media.

Homogenized tissue samples were placed in broth with thioglycollate medium. The cultures were incubated at 37°C for up to 14 days, subcultured on solid nutrient media: on the 1st day - on Columbia, Chocolate and Schedler agars; on the 5th day - on Chocolate and Schedler agar and on the 10th day - only on Schedler agar. For aerobic, anaerobic and capnophilic microorganisms, incubation conditions were created using gas-generating packages.

Identification of isolated microorganisms and sensitivity to antibiotics was carried out using an automatic analyzer (Vitec2 compact; Bio Merieux, France) and a semi-automatic analyzer (Multiscan FC; Thermo Fisher, USA) using kits (Erba Lachema, Czech Republic), test systems ("Diagnostic systems", Russia).

Sensitivity to antibacterial drugs was tested using the disk diffusion method and analyzer kits. Antibiotic sensitivity assessment was carried out in accordance with the criteria of EUCAST 2018 (studies in 2018-2019), EUCAST 2021 (studies in 2021-2022).

ELIGIBILITY:
Inclusion Criteria:

* Clinically confirmed periprosthetic infection

Exclusion Criteria:

* No signs of periprosthetic infection

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The sample included cases of deep and superficial infection after arthroplasty of the knee, hip, shoulder and wrist joints, regardless of the location of the primary operation. Isolated microorganisms were identified based on growth in one or more cultures obtained from punctate synovial fluid, intraoperative tissues, and from removed implants (after their ultrasonic treatment).
Sampling Method: Non-Probability Sample
Enrollment: 342 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Structure of isolated pathogens of periprosthetic infection | 2018-2019
  The proportion of identified microorganisms in the general structure of pathogens of periprosthetic infection
Structure of isolated pathogens of periprosthetic infection | 2021-2022
  The proportion of identified microorganisms in the general structure of pathogens of periprosthetic infection

SECONDARY OUTCOMES:
Antibiotic resistance of isolated pathogens of periprosthetic infection | 2018-2019
  Sensitivity to antibacterial drugs was tested using the disk diffusion method and analyzer kits. Antibiotic sensitivity assessment was carried out in accordance with the criteria of EUCAST 2018 (studies in 2018-2019).
Antibiotic resistance of isolated pathogens of periprosthetic infection | 2021-2022
  Sensitivity to antibacterial drugs was tested using the disk diffusion method and analyzer kits. Antibiotic sensitivity assessment was carried out in accordance with the criteria of EUCAST 2021 (studies in 2021-2022).

CONTACTS AND LOCATIONS:
Locations (1):
- Federal Center for Traumatology, Orthopedics and Endoprosthetics, Cheboksary, Chuvashskaya Respublika, Russia

IPD SHARING:
Plan to Share IPD: Undecided
On request